CLINICAL TRIAL: NCT00661258
Title: Antiretroviral Treatment Adherence for Life Pilot Study: Phases II and III
Brief Title: China Antiretroviral Treatment Adherence for Life
Acronym: AFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Beijing Ditan Hospital (Other); Second People's Hospital, Dali (Other)
Responsible Party: Principal Investigator, Lora Sabin, Associate Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25495; GHS-A-00-03-00030-00 (Other Grant/Funding Number: GHS-A-00-03-00030-00)
Record Dates: First submitted 2008-04-11; First posted 2008-04-18 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections
Keywords: HIV antiretroviral treatment adherence intervention China; adherence to antiretroviral treatment; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group patients were given their electronic drug monitoring feedback data at each monthly visit. The study coordinator would quickly calculate whether the patient's adherence was below 95% in the previous month. If so, that patient was flagged for enhanced counseling with a clinic doctor and this counseling was based on a printout containing the electronic drug monitoring data.
  Interventions: Behavioral: Electronic drug monitoring feedback data
- Comparison (No Intervention): The comparison group patients were not given the data from the electronic data monitoring feedback data. Instead, they filled out a self report form that all patients fill out. If they indicated in this report that their adherence in the previous was less than 95%, then they were flagged for "enhanced counseling" with a doctor. This counseling was based on the patient's self report. Thus both groups received enhanced counseling if they indicated poor adherence, but only the intervention group were given their electronic data output.

INTERVENTIONS:
Behavioral: Electronic drug monitoring feedback data — All patients were given electronic drug monitors that can monitor pill-taking behavior. In the intervention arm, patients and their attending doctors were given the electronic drug monitoring data on pill bottle openings at each monthly visit for use in adherence counseling sessions. Control arm patients were not given their electronic drug monitoring feedback data and their counseling sessions were based on self-reported adherence, as per standard of care in Dali.
  Arms: Intervention

SUMMARY:
This study focuses on collecting and analyzing quantitative data related to adherence to antiretroviral treatment from patients in Dali, China, over a one-year time-frame and generating preliminary data on an intervention designed to improve adherence to antiretroviral treatment among the study population.

DETAILED DESCRIPTION:
This study is a continuation of "Adherence for Life (AFL): Phase I: Exploratory Research" (H-25203), which focused on collecting and analyzing qualitative data on adherence to antiretroviral treatment (ART) among HIV-positive patients in Dali, Yunnan Province, China. Like Phase I, the AFL Pilot Study (Phases II and III) will be a collaborative effort between US researchers based in Boston, MA and Chinese researchers based in Beijing and Dali. The current study, Phases II and III, will focus on collecting and analyzing qualitative and quantitative data related to adherence to ART over a one-year time-frame and generating preliminary data on an intervention designed to improve adherence to ART among the study population. The questionnaires used in these phases of the study will draw on the results of Phase I as well as standardized instruments adapted to the Chinese context. The specific aims of the study are as follows: (1) To determine the best surrogate measure of ART adherence among the study population; (2) To determine ART adherence rates in this population; (3) To analyze the relationship between adherence factors and measured adherence rates; and (4) To generate preliminary effectiveness data on an intervention that makes use of electronic drug monitors (EDM) to improve ART adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older, currently on antiretroviral treatment or about to begin it, live in the study catchment area, and are willing to provide informed consent.

Exclusion Criteria:

* Persons below the age of 18 years, persons who are not currently on or about to start antiretroviral treatment, persons who live outside the study catchment area, or person not willing to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora L Sabin, PhD, Principal Investigator — Center for International Health and Development, Boston University
Locations (1):
- Dali Second People's Hospital, Dali, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 patients were recruited at the Dali 2nd People's Hospital, in Dali, Yunnan Province, from June to November 2006 in the 6-month pre-intervention period. A total of 68 patients completed this passive phase and were randomized to intervention vs. control arm.
Groups:
- Intervention: The intervention group patients were given their electronic drug monitoring data at each monthly visit. The study coordinator would quickly calculate whether the patient's adherence was below 95% in the previous month. If so, that patient was flagged for enhanced counseling with a clinic doctor and this counseling was based on a printout containing the electronic drug monitoring data.
- Control: The control group patients were not given the data from the electronic data monitoring. Instead, they filled out a self report form that all patients fill out. If they indicated in this report that their adherence in the previous was less than 95%, then they were flagged for "enhanced counseling" with a doctor. This counseling was based on the patient's self report. Thus both groups received enhanced counseling if they indicated poor adherence, but only the intervention group were given their electronic data output.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 34 | 34
Completed | 31 | 33
Not Completed | 3 | 1
Not completed — Death | 1 | 0
Not completed — caught by police and in detox center | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (8.3) | 35.1 (8.0) | 35.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  China | 34 | 34 | 68

OUTCOME MEASURES:

1. Secondary Outcome: Change in CD4 Count
Description: Mean change in CD4 count (cells/µL) between Month 6 and Month 12 (pre-intervention vs. last month of intervention)
Time Frame: Month 6, Month 12
Measure: Mean (Standard Deviation); unit: cells/µL
Groups:
- Control: The control group patients were not given the data from the electronic data monitoring. Instead, they filled out a self report form that all patients fill out. If they indicated in this report that their adherence in the previous was less than 95%, then they were flagged for
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 33
cells/µL | 90.0 (171.6) | -8.8 (152.6)

2. Primary Outcome: Mean Adherence, as Measured by Electronic Drug Monitors (EDM)
Description: We used the electronic drug monitors (EDM) adherence metric that was found to be most strongly associated with viral suppression (HIV RNA <400 copies/ml) in analysis of the pre-intervention data, EDM 'proportion taken within dose time' (see Gill et al, 2009). This measure estimated monthly adherence as the proportion of prescribed doses taken on time, e.g., within 1 hour of scheduled dose time ([number of doses taken ±1 hour of dose time] / [total number of prescribed doses]).
Time Frame: Month 12 (last month of 6-month intervention period) and 6-month post-intervention period
Population: Of 68 subjects randomized at 6 months, 64 completed the full 12 months of data collection, 31 in Intervention Arm and 33 in Comparison Arm.
Measure: Mean (Standard Deviation); unit: percentage of doses taken on time
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 33
percentage of doses taken on time
  Mean adherence in Month 12 | 96.5 (4.8) | 84.5 (21.0)
  Mean adherence in intervention period (Months 7-12 | 96.4 (3.4) | 84.1 (21.4)

ADVERSE EVENTS:
Time Frame: 1 year of data collection
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No